CLINICAL TRIAL: NCT04257019
Title: Assessing the Effect of Lavender on Pain and Anxiety Levels During Interventional Spine Procedures Under Fluoroscopy
Brief Title: Pain, Anxiety During Interventional Spine Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Chong Kim, PI, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB19-00512
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pain; Low Back Pain; Procedural Pain; Procedural Anxiety
Keywords: lavender; procedural pain; patient experience
MeSH Terms: conditions — Pain; Low Back Pain; Pain, Procedural | interventions — lavender oil; almond oil; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lavender (Experimental): Lavender mask before and during procedure
  Interventions: Other: Lavender oil
- Almond (Active Comparator): Almond oil mask before and during procedure
  Interventions: Other: Almond oil
- Water (Sham Comparator): Water mask before and during procedure
  Interventions: Other: Water

INTERVENTIONS:
Other: Lavender oil — Inhalation of Lavender oil
  Arms: Lavender
Other: Almond oil — Inhalation of Almond oil
  Arms: Almond
Other: Water — Inhalation of water
  Arms: Water

SUMMARY:
Lavender is a plant whose extracts are widely used in aromatherapy. Lavender has been shown to decrease pain during procedures, and has also been shown to decrease pre-operative anxiety. It contains two compounds, linalool and linalyl acetate, both of which have been shown to stimulate the parasympathetic nervous system. The study will be conducted to evaluate the effect of inhaled lavender on pain and anxiety levels associated with specific interventional pain procedures. The study will be conducted in a randomized controlled trial. The trial will include one experimental group who will be exposed to lavender oil infused surgical mask to be worn by the subject, a second placebo group who will be exposed to a almond oil infused surgical mask to be worn, and a third control group who will wear a surgical mask infused with sterile water. Participants will be randomly assigned, and subject will be blinded. Our study will seek at least sixty participants, each randomly assigned either the experimental, placebo, or control group (n=20) to ensure adequate power. The disease characteristics among groups will be similar, with all participants experiencing back pain with or without radicular symptoms leading them to seek lumbar epidural steroid injection or lumbar medial branch block. Pre-procedural anxiety and anxiety occurring during the procedure will be measured by the State Trait Anxiety Inventory (STAT-I) questionnaire. Procedural pain will be measured using the Visual Analogue Scale (VAS). Our goal with this study is to investigate safe, adjunctive therapies that may decrease patient discomfort during interventional pain procedures, and ultimately improve procedural adherence.

DETAILED DESCRIPTION:
Interventional spine procedures such as lumbar epidural steroid injections and nerve blocks can be painful or anxiety provoking for patients. It is paramount to reduce pain and anxiety as much as possible during these procedures, since doing so improves patient satisfaction and compliance.

Lavender is a plant whose extracts are widely used in aromatherapy. Aromatherapy is defined as the therapeutic use of essential oils derived from plants. Lavender aromatherapy has been reported to possess several therapeutic effects including anti-anxiety, sedation, mood stabilization, and analgesia.

Situational anxiety, such as that relating to procedures, along with procedural pain, can be particularly uncomfortable for patients. The current short-acting anxiolytic agents like benzodiazepines and pain-relieving opiates are associated with numerous side effects such as drug tolerance, abuse and sedation. Consequently, it is important to discover an alternative therapy to relieve anxiety and pain. Lavender has been shown to decrease anxiety in patients scheduled to undergo colorectal surgery and has been shown to decrease anxiety associated with dental procedures. Lavender has also been shown to decrease pain during procedures, particularly when inhaled prior to a generally painful procedure such as catheter or needle insertion, or chest tube removal.

Two basic mechanisms may explain the effects of lavender therapy. First is the influence of aroma on the brain through the limbic system via olfaction, and the other is through the direct pharmacological effects of the essential oil. Lavender contains two compounds, linalool and linalyl acetate, both of which have been shown to stimulate the parasympathetic nervous system. In recent animal models, linalyl acetate anxiolytic effects were not observed in anosmic mice, indicating that the effects were triggered by olfactory input. In addition, it was found that flumazenil antagonized odor-induced anxiolytic effects, indicating that GABAergic transmission plays an important role in anxiolytic effects.

It is well known that anxiety can alter the course of pain. Studies show that the emotional and behavioral responses to pain are strongly guided by two related psychosocial factors, fear and anxiety. Individuals who have lower anxiety do not interpret pain as negatively, which aids in recovery.

This study seeks to investigate whether lavender essential oil reduces pain and anxiety during interventional spine procedures.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are undergoing lumbar epidural steroid injections or lumbar medial branch blocks
2. Age 21 or older

Exclusion Criteria:

1. An allergy or sensitivity to lavender or almond oil
2. A pre-existing problem with the sense of smell
3. A subject unable to follow basic instructions relating to the design of the experiment, or subjects unable to answer questions regarding their pain or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Pain perception | 1 day
  Perception of pain, VAS

SECONDARY OUTCOMES:
Anxiety | 1 day
  Anxiety related to procedure

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided